CLINICAL TRIAL: NCT06328530
Title: Repetitive Applications of Pruritogens and Effects of a Cutaneous-induced Pain Stimulation on Nonhistaminergic Itch Perception
Brief Title: Itch Sensation Induced by Simultaneous Application of Pruritogens (Spatial Summation)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate Professor, Aalborg University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20210046 3rd project
Record Dates: First submitted 2024-03-19; First posted 2024-03-25 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Histamine; Cowhage
MeSH Terms: interventions — Histamine

STUDY DESIGN:
Intervention Model Description: The participants will randomly receive applications of cowhage and histamine.
Who Masked: Participant
Masking Description: Participant will be blinded about application of pruritogens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st pruritogen (Experimental): The subproject consists of 2 sessions 3 days apart. Each session consists of 3 parts.
  In the first session, 3 test areas (4x4 cm) will be selected on the subject's forearms. In part 1, we will apply cowhage in one area. In part 2, we will apply cowhage in two areas on the same arm. In part 3, we will again apply cowhage in 2 areas, one on each arm. In each part, the itch intensity will be measured using a VAS (visual analog scale) for 10 min from the cowhage application. After removal of the cowhage, alloknesis and mechanically evoked itch will be measured in the area selected in part 1.
  Interventions: Other: Cowhage
- 2nd pruritogen (Other): The second session will take place 3 days after the first one and will follow the same procedure as session 1. However, histamine will be applied instead of cowhage. The order of the two sessions will be randomized.
  Interventions: Other: Histamine

INTERVENTIONS:
Other: Cowhage — 25 spicules will be inserted in the center of the predefined skin area on the mandibular area. The spicules will be gently rubbed for 15-20 seconds in circular motion to facilitate epidermal penetration.
  Arms: 1st pruritogen
Other: Histamine — Histaminergic itch will be evoked by a 1% histamine solution. A droplet of histamine solution will be placed on the predetermined area on the forearm, and the SPT lancet will be pierced through the histamine with 120 g of pressure for 1-2 seconds.
  Arms: 2nd pruritogen

SUMMARY:
In This experiment, the investigators would like to design a new itch model based on the spatial summation of pruritic stimuli. The hypothesis behind this study (spatial summation) is that two simultaneous applications of pruritogens will result in higher itch sensation compared with a single application of pruritogen.

DETAILED DESCRIPTION:
Chronic itch affects approximately a fifth of the global population and is associated with substantial negative consequences for the affected individuals. Furthermore, there is a lack of efficient treatment options for chronic itch. In order to mimic a clinical itch condition as presented in patients, the aim of the project is to investigate a new itch model based on the spatial summation of pruritic stimuli. The aim of this experiment is to assess the itch sensation induced by simultaneous application of pruritogens (spatial summation). In particular, the purpose is to evaluate if a single application of cowhage/histamine (non-histaminergic and histaminergic itch respectively) results in a lower itch sensation compared to two simultaneous applications of the pruritogens, on the same arm or in different arms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other addictive drugs
* Previous or current history of neurological (e.g. neuropathy), immunological (e.g. asthma, immune deficiencies, arthritis) musculoskeletal (e.g. muscular pain in the upper extremities,), cardiac disorder, or mental illnesses that may affect the results
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics, and pain killers, as well as systemic or topical steroids
* Skin diseases (e.g. atopic dermatitis, pruritus nodularis, eczema, psoriasis)
* Moles, scars, or tattoos in the area to be treated or tested.
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of itch | 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the itch intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no itch' and 100 'worst itch imaginable'.
Assessment of pain | 1 minute after every itch inductions
  Immediately following the itch provocations, participants will be instructed to rate the pain intensity for 10 minutes using a digital visual analogue scale (VAS; eVAS Software: Aalborg, University, Denmark), on a tablet. The scale will be measured from 0 to 100, where 0 represents 'no pain' and 100 'worst pain imaginable'.

SECONDARY OUTCOMES:
Alloknesis | 12 minutes after every itch inductions
  Alloknesis sensation is measured using a standardized sensory brush (SENSELab Brush-05, Somedic AB, Hörby, Sweden) exerting a force of 200 to 400 mN.
Mechanically evoked itch | 15 minutes after every itch inductions
  Mechanically evoked itch is measured using three von Frey filaments of 4.08, 4.16 and 4.31 (1.0, 1.4, 2.0 g, respectively) (North Coast Medical, Gilroy, CA). The center of the skin area is stimulated by 3 pricks, repeated 3 times in short succession. After a total of 9 stimulations, the participants will report the itch elicited on a numerical rating scale (NRS) from 0 to 10 (0 = "no itch"; 10 = "worst imaginable itch").

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark